CLINICAL TRIAL: NCT05141825
Title: Proton and Carbon Ion Radiotherapy for Cervical Cancer : A Retrospective Analysis
Brief Title: Proton and Carbon Ion Radiotherapy for Cervical Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shanghai Proton and Heavy Ion Center (Other)
Responsible Party: Principal Investigator, Zhan Yu, physician of abdorminal and pelvic oncology department, Shanghai Proton and Heavy Ion Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPHIC-TR-CERC-2021-01
Record Dates: First submitted 2021-11-23; First posted 2021-12-02 (Actual); Last update posted 2021-12-02 (Actual); Status verified 2021-11

CONDITIONS: Cervical Cancer
Keywords: proton and carbon ion radiotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Protons; Heavy Ion Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- proton and carbon ion radiotherapy (Experimental): proton and carbon ion radiotherapy
  Interventions: Radiation: proton and carbon ion radiotherapy

INTERVENTIONS:
Radiation: proton and carbon ion radiotherapy — proton and carbon ion radiotherapy

SUMMARY:
The aim of this study is to evaluate the toxicity and tolerance of proton and carbon ion radiotherapy (PCRT) for cervical cancer.

DETAILED DESCRIPTION:
To retrospectively analyze cervical cancer patients received radical proton and carbon radiotherapy in our center. The acute and late toxicities, overall survival (OS), local control rate (LC), progression-free survival (PFS) and distant metastasis-free survival (DMFS) were analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. . histologically diagnosis of squamous cell carcinoma of the cervix;
2. . International Federation of Gynecology and Obstetrics (FIGO) stage (2014) IB2 - IIIB, without rectum invasion; or FIGO stage IA - IB1, who refused surgery or were contraindication for surgery due to comorbidity diseases;
3. . received proton and carbon ion radiotherapy (PCRT) with or without chemotherapy for curative intention;
4. . Follow-up data available.

Exclusion Criteria:

1. a previous history of other malignancy;
2. squamous cell carcinoma of the cervix patients who had received surgery;
3. rectum was invaded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | through study completion, an average of 1 year
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

SECONDARY OUTCOMES:
overall survival rate | 3 years
  overall survival rate
local control rate | 3 years
  local control rate
progression-free survival | 3 years
  progression-free survival
distant metastasis-free survival | 3 years
  distant metastasis-free survival

CONTACTS AND LOCATIONS:
Overall Officials: Qing Zhang, MD, Principal Investigator — Shanghai Proton and Heavy Ion Center

IPD SHARING:
Plan to Share IPD: No